CLINICAL TRIAL: NCT00645866
Title: A Neo-Adjuvant Study of Sequential Epirubicin and Docetaxel in Combination With Capecitabine in Patients With Locally Advanced Breast Cancer
Brief Title: Epirubicin, Docetaxel, and Capecitabine in Treating Women With Stage IIIA or Stage IIIB Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Julian R. Molina, M.D., Ph.D., Mayo Clinic Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582618; P30CA015083 (NIH); MC0132 (Other: Mayo Clinic Cancer Center); 595-02 (Other: Mayo Clinic IRB); 378-ONC-0030-241 (Other: Pharmacia Protocol)
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel; Epirubicin; Pharmacogenomic Testing; Biopsy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: docetaxel
Drug: epirubicin hydrochloride
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Procedure: biopsy
Procedure: neoadjuvant therapy
Procedure: therapeutic surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, docetaxel, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving epirubicin together with docetaxel and capecitabine and to see how well it works in treating women with stage IIIA or stage IIIB breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Describe the pathologic response rate in chemotherapy-naive women with locally advanced breast cancer (stage IIIA or IIIB) after 6 courses of sequential neoadjuvant therapy with epirubicin hydrochloride and a combination of docetaxel with capecitabine .
* Describe the adverse events of sequential epirubicin hydrochloride and a combination of docetaxel with capecitabine in this patient population.

Secondary

* Identify by transcriptional profiling the differential expression of candidate gene products that confer chemosensitivity to epirubicin hydrochloride, docetaxel, and capecitabine.
* Correlate the differential expression of known genetic polymorphisms of intracellular regulators involved in the metabolism of epirubicin hydrochloride, docetaxel, and capecitabine with adverse events and tumor response.
* Assess individual patient variation in clinical (toxicity and/or activity), in pharmacologic (pharmacokinetic/pharmacodynamic parameters), and/or biologic (correlative laboratory study results) responses to epirubicin hydrochloride, docetaxel, and capecitabine due to genetic differences in proteins involved in drug response (transport, metabolism and/or mechanism of action).

OUTLINE: Patients receive epirubicin hydrochloride IV on day 1. Treatment repeats every 2 weeks for 3 courses. Beginning 2 weeks after last dose of epirubicin hydrochloride, patients receive docetaxel IV over 1 hour on day 1 and oral capecitabine twice daily on days 1-14. Treatment with docetaxel and capecitabine repeats every 3 weeks for 3 courses. Patients then undergo surgery.

Blood samples are collected at baseline for pharmacogenetic studies. Tumor tissue samples are collected at baseline and periodically during treatment for correlative laboratory studies.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Stage IIIA or IIIB disease (T3 N1 M0, T4 N1 M0, any T N2/N3 M0)
* Bidimensionally measurable or evaluable disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Platelet count ≥ 100,000 cells/μL
* Total bilirubin normal
* Hemoglobin ≥ 8.0 g/dL
* ANC ≥ 1,000 cells/μL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine clearance ≥ 50 mL/min and serum creatinine normal
* Life expectancy ≥ 3 months
* No uncontrolled infection
* No chronic debilitating disease
* No lack of physical integrity of the upper gastrointestinal tract
* Able to swallow tablets
* No malabsorption syndrome
* No clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias [New York Heart Association class III-IV heart disease] or myocardial infarction within the last 12 months)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer or adequately treated other noninvasive carcinomas
* No peripheral neuropathy ≥ grade 1

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior major surgery and recovered
* No prior chemotherapy regimens including adjuvant therapy
* No organ allograft
* No concurrent sorivudine or bruvidine
* No other concurrent cytostatic, cytotoxic, immunomodulating agents, or radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2003-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Pathologic response rate
Toxicity patterns

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Julian R. Molina, MD, PhD, Study Chair — Mayo Clinic; James N. Ingle, MD, Principal Investigator — Mayo Clinic; Wilma Lingle, PhD, Principal Investigator — Mayo Clinic